CLINICAL TRIAL: NCT05133817
Title: Prophylactic Norepinephrine Infusion Combined With 6% Hydroxyethyl Starch (130/0.4) Coload for Postspinal Anesthesia Hypotension in Patients Undergoing Cesarean Section: A Randomized, Controlled, Dose-finding Trial
Brief Title: Prophylactic Norepinephrine Infusion Combined With Colloid Coloading for Postspinal Anesthesia Hypotension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Yi Chen-2021-5
Record Dates: First submitted 2021-11-12; First posted 2021-11-24 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2021-11

CONDITIONS: Adverse Event
Keywords: Norepinephrine; Hydroxyethyl starch; Postspinal anesthesia hypotension; Coload; Cesarean section
MeSH Terms: interventions — Saline Solution; Norepinephrine; Vasoconstrictor Agents

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control group (Placebo Comparator): Simultaneous with spinal anesthesia, 500 mL 6% Hydroxyethyl starch (130/0.4) coload was given and a maintenance dose of normal saline by IV infusion.
  Interventions: Drug: Normal saline
- 0.025 μg/kg/min group (Experimental): Simultaneous with spinal anesthesia, 500 mL 6% Hydroxyethyl starch (130/0.4) coload was given and a maintenance dose of norepinephrine (0.025 μg/kg/min) by IV infusion.
  Interventions: Drug: Norepinephrine (0.025 μg/kg/min)
- 0.05 μg/kg/min group (Experimental): Simultaneous with spinal anesthesia, 500 mL 6% Hydroxyethyl starch (130/0.4) coload was given and a maintenance dose of norepinephrine (0.05 μg/kg/min) by IV infusion.
  Interventions: Drug: Norepinephrine (0.05 μg/kg/min)
- 0.075 μg/kg/min group (Experimental): Simultaneous with spinal anesthesia, 500 mL 6% Hydroxyethyl starch (130/0.4) coload was given and a maintenance dose of norepinephrine (0.075 μg/kg/min) by IV infusion.
  Interventions: Drug: Norepinephrine (0.075 μg/kg/min)
- 0.1μg/kg/min group (Experimental): Simultaneous with spinal anesthesia, 500 mL 6% Hydroxyethyl starch (130/0.4) coload was given and a maintenance dose of norepinephrine (0.1μg/kg/min) by IV infusion.
  Interventions: Drug: Norepinephrine (0.1 μg/kg/min)

INTERVENTIONS:
Drug: Normal saline — Simultaneous with spinal anesthesia, 500 mL 6% Hydroxyethyl starch (130/0.4) coload was given and a maintenance dose of normal saline by IV infusion.
  Other Names: NS
  Arms: Control group
Drug: Norepinephrine (0.025 μg/kg/min) — Simultaneous with spinal anesthesia, 500 mL 6% Hydroxyethyl starch (130/0.4) coload was given and a different maintenance dose of norepinephrine by IV infusion.
  Other Names: Vasopressor
  Arms: 0.025 μg/kg/min group
Drug: Norepinephrine (0.05 μg/kg/min) — Simultaneous with spinal anesthesia, 500 mL 6% Hydroxyethyl starch (130/0.4) coload was given and a different maintenance dose of norepinephrine by IV infusion.
  Other Names: Vasopressor
  Arms: 0.05 μg/kg/min group
Drug: Norepinephrine (0.075 μg/kg/min) — Simultaneous with spinal anesthesia, 500 mL 6% Hydroxyethyl starch (130/0.4) coload was given and a different maintenance dose of norepinephrine by IV infusion.
  Other Names: Vasopressor
  Arms: 0.075 μg/kg/min group
Drug: Norepinephrine (0.1 μg/kg/min) — Simultaneous with spinal anesthesia, 500 mL 6% Hydroxyethyl starch (130/0.4) coload was given and a different maintenance dose of norepinephrine by IV infusion.
  Other Names: Vasopressor
  Arms: 0.1μg/kg/min group

SUMMARY:
The purpose of this study is to investigate the suitable infusion dose of prophylactic norepinephrine infusion combined with 6% Hydroxyethyl starch (130/0.4) coload for post-spinal anesthesia hypotension in patients undergoing cesarean section.

DETAILED DESCRIPTION:
Post-spinal anesthesia hypotension is a frequent complication during spinal anesthesia for cesarean section. The incidence of post-spinal anesthesia hypotension is as high as 62.1-89.7% if prophylactic measures are not taken. Vasopressor has been highly recommended for routine prevention and/or treatment of post-spinal anesthesia hypotension. As a potential substitute drug for phenylephrine, norepinephrine has gradually been used in parturients undergoing cesarean section. There's some evidence that prophylactic infusion of norepinephrine could effectively reduce the incidence of post-spinal anesthesia hypotension in parturients undergoing cesarean section. But the ideal infusion dose of norepinephrine with colloid coload is still unknown. The purpose of this study is to investigate the suitable infusion dose of prophylactic norepinephrine infusion combined with 6% Hydroxyethyl starch (130/0.4) coload for post-spinal anesthesia hypotension in patients undergoing cesarean section.

ELIGIBILITY:
Criteria: Inclusion Criteria:

* 18-40 years
* Primipara or multipara
* Singleton pregnancy ≥ 37 weeks
* American Society of Anesthesiologists physical status classification I to II
* Scheduled for elective cesarean section under spinal anesthesia

Exclusion Criteria:

* Body height < 150 cm
* Body weight > 100 kg or body mass index (BMI) ≥ 40 kg/m2
* Eclampsia or chronic hypertension or baseline blood pressure ≥ 160mmHg
* Hemoglobin < 7g/dl
* Coagulation or renal function disorders
* Known allergy to hydroxyethyl starch
* Fetal distress, or known fetal developmental anomaly

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 175 (Actual)
Dates: Start 2021-11-26 (Actual); Primary Completion 2022-09-03 (Actual); Study Completion 2022-09-03 (Actual)

PRIMARY OUTCOMES:
The incidence of post-spinal anesthesia hypotension | 1-15 minutes after spinal anesthesia
  Systolic blood pressure (SBP) < 80% of the baseline

SECONDARY OUTCOMES:
Overall stability of systolic blood pressure control versus baseline | 1-15 minutes after spinal anesthesia
  Evaluated by performance error (PE).
The incidence of severe post-spinal anesthesia hypotension. | 1-15 minutes after spinal anesthesia
  Systolic blood pressure (SBP) < 60% of the baseline.
The incidence of nausea and vomiting. | 1-15 minutes after spinal anesthesia
  Presence of nausea and vomiting in patients after spinal anesthesia
The incidence of bradycardia. | 1-15 minutes after spinal anesthesia
  Heart rate < 55 beats/min.
The incidence of hypertension. | 1-15 minutes after spinal anesthesia
  Systolic blood pressure (SBP) >120% of the baseline.
pH value | Immediately after fetal delivery
  Analyse from umbilical arterial blood gases.
Partial pressure of oxygen | Immediately after fetal delivery
  Analyse from umbilical arterial blood gases.
Concentration of base excess | Immediately after fetal delivery
  Analyse from umbilical arterial blood gases.
Apgar score (0-10; a higher score means a better outcome) | 5 min after fetal delivery
  A= Appearance (0-2); P=Pulse (0-2); G=Grimace (0-2); A=Attitude (0-2); R=Respiration (0-2)
Apgar score (0-10;a higher score means a better outcome) | 5 min after fetal delivery
  A= Appearance (0-2); P=Pulse (0-2); G=Grimace (0-2); A=Attitude (0-2); R=Respiration (0-2)

CONTACTS AND LOCATIONS:
Overall Officials: Yi Chen, M.D., Study Chair — General Hospital of Ningxia Medical University
Locations (1):
- General Hospital of Ningxia Medical University, Yinchuan, Ningxia, China

REFERENCES:
- [Derived] Guo L, Xiong X, Qin R, Li Z, Shi Y, Xue W, He L, Ma S, Chen Y. Prophylactic norepinephrine combined with 6% hydroxyethyl starch (130/0.4) co-load infusion for preventing postspinal anesthesia hypotension during cesarean section: a randomized, controlled, dose-finding trial. Daru. 2024 Jun;32(1):1-9. doi: 10.1007/s40199-023-00479-7. Epub 2023 Oct 9. PMID 37812381